CLINICAL TRIAL: NCT03589742
Title: Feasibility Study for Optically Guided Radiofrequency Ablation Catheter
Acronym: NEOVIEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medlumics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-001890-34; 2016-001890-34 (EudraCT Number)
Record Dates: First submitted 2018-06-22; First posted 2018-07-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Radiofrequency Ablation; Pulmonary Vein Isolation; Catheter; AblaView Ablation Catheter; Atrioventricular node
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency ablation patients (Experimental): Single-Arm study, all patients included will undergo RF ablation using AblaView® Ablation Catheter
  Interventions: Device: AblaView® Ablation Catheter

INTERVENTIONS:
Device: AblaView® Ablation Catheter — The AblaView® Ablation Catheter is a regular RF ablation catheter with the same physical characteristics and the same biocompatible materials, with an 8 French (2.66 mm) sheath and 180º deflection angle. The tip of the catheter has 15 holes distributed around it where the irrigation will be delivered into the patient's blood. The front irrigation hole will deliver at the same time the infrared light for the OCR system.

SUMMARY:
Clinical study intended to evaluate the feasibility of a new irrigated RF ablation catheter that allows the physiologist to perform a regular RF ablation procedure while it is being monitored through an imaging technique known as Optical Coherence Reflectometry (OCR). This technique is based upon the use of infrared light; it is innocuous for the human body and allows for the detection of the contact between the catheter tip with the tissue besides the lesion formation during the Radiofrequency (RF) application as the OCR technique is able to distinguish between ablated tissue and healthy tissue. Both features are able to provide a better control of the ablation procedure, which may become in a better clinical result in cardiac ablation procedures, especially in Atrial Fibrillation cases.

DETAILED DESCRIPTION:
This feasibility study intended for the evaluation of the technique in humans prior to a Safety and efficacy study based on the non-inferiority of AblaView® Ablation Catheter against a control device. Thus, no randomization has been decided and no blinding has been considered necessary.

The primary clinical endpoints of this investigation are as follows:

* Primary Endpoint 1: Feasibility of the technique in humans. Validate that the technique is able to provide real time image of the change in the optical properties of the heart tissue during the ablation procedure.
* Primary Endpoint 2: Safety of the technique, major complications incidence (equal to or below regular procedure incidence of serious adverse events of 5%) 30 days after the procedure (ictus, cardiac tamponade, major hemorrhage, esophageal lesion, death)
* Secondary Endpoint 1: Safety of the device, complications incidence within the 30 days after the procedure (Detachable parts, irrigation leak, malfunction of the handling/steering, break of electrical parts and "pop" occurrence) The Principal Investigator will be responsible for the evaluation of the Primary Endpoint 1, providing feedback from every patient and describing the feasibility of the technique according to his criteria.

The Primary Endpoint 2 will be measured according to the clinical practice guidance for the evaluation of: ictus, cardiac tamponades, major hemorrhage, esophageal lesion and death, and will be recorded right after the procedure and in the patient record for the 30 days follow up visit.

The Secondary Endpoint 1 will be measured according to the Principal investigator's criteria and the assessment of the Medlumics technician for the evaluation of detachable parts, irrigation leaks, malfunction of the handling/steering, break of electrical parts and "pop" occurrence), and will be recorded right after the procedure and in the patient record for the 30 days follow up visit.

Subjects will only be replaced if the recruitment period is not ended and the eligible number of patients is under 15, they will not be replaced if they get excluded after the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients with confirmed paroxysmal Atrial Fibrillation, showing symptoms, with a documented episode within the last year, where at least 1 antiarrhythmic drug treatment have failed, and considered as candidates for cardiac ablation after electrophysiologist diagnose
* Patients with confirmed Atrial Flutter, showing symptoms, with a documented episode within the last year, and considered as candidates for cardiac ablation after electrophysiologist diagnose
* All patients will be properly informed, accepting to participate in the study voluntarily by signing the informed consent form.

Exclusion Criteria:

* Patients that have been subject of a former RF ablation procedure weather for Atrial Fibrillation or Atrial Flutter
* Patients with significant structural cardiopathy (ventricular dysfunction with Left Ventricle Ejection Fraction (LVEF)<35%, with severe valvulopathies, congenital cardiopathies)
* Severe dilatation of the left atria (>5 cm)
* Acute coronary syndrome within the last year prior to enrolment
* Any hemorrhagic ictus or ischemic ictus within the last year prior to enrolment
* Active hemorrhage
* Anticoagulant contraindications
* Patients with severe comorbidities that may reduce their life expectancy (<1 year) or personal circumstances that may difficult the clinical follow up
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of the technique in humans | at completion of the procedure with AblaView® Ablation Catheter
  Validate that the technique is able to provide real time image of the change in the optical properties of the heart tissue during the ablation procedure. This change will be analyzed intraoperative because untreated myocardial tissue has a high level of cellular organization, which exhibits a significant phase retardation between orthogonal polarization states, leading to reflect polarized light. But birefringence property disappears by applying RF power during time on the same location, because the fibers are denaturalized. This optical change can be measured to provide a reliable marker for cellular and subcellular organization to estimate lesion formation in real time

SECONDARY OUTCOMES:
Incidence of the technique on occurence of adverse effects (Safety and Tolerability) | 30 days after the procedure
  major complications incidence (equal to or below regular procedure incidence of serious adverse events of 5%) within the 30 days after the procedure (ictus, cardiac tamponade, major hemorrhage, esophageal lesion, death)
Validation of the usability and design of the medical device | 30 days after the procedure of ablation with AblaView® Ablation Catheter is completed
  complications incidence within the 30 days after the procedure (Detachable parts, irrigation leak, malfunction of the handling/steering, break of electrical parts and "pop" occurrence)

CONTACTS AND LOCATIONS:
Overall Officials: Stepan Kralovec, Study Director — Authorised representative in the Czech Republic; Petr Neuzil, MD, Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herranz D, Lloret J, Jimenez-Valero S, Rubio-Guivernau JL, Margallo-Balbas E. Novel catheter enabling simultaneous radiofrequency ablation and optical coherence reflectometry. Biomed Opt Express. 2015 Aug 7;6(9):3268-75. doi: 10.1364/BOE.6.003268. eCollection 2015 Sep 1. PMID 26417499